CLINICAL TRIAL: NCT00663793
Title: Oral Androgens in Man-6: Pharmacokinetics of Slow and Fast Release, External Matrix Oral Testosterone Formulations in Normal Men With Experimental Hypogonadism
Brief Title: ORAL T-6: Oral Androgens in Man-6
Acronym: ORAL-T-6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33738-B; U54HD42456-06 (Other Grant/Funding Number: NIH/NICHD); K23HD045386 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-12

CONDITIONS: Contraception; Hypogonadism
Keywords: Male Contraception; Hypogonadism; Testosterone
MeSH Terms: conditions — Hypogonadism | interventions — acyline; Testosterone; Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral testosterone (Experimental): (Day 1) Acyline 300 mcg/kg once, followed 24 hours later (Day 2) by "immediate release" T 300 mg po once (as a control), followed 24 hours later (Day 3) by "external matrix fast release" T 300 mg once, followed 24 hours later (Day 4) by "external matrix slow release" T 300 mg once, followed 96 hours later (Day 8) by "immediate release" T 600 mg, followed 24 hours later (Day 9) by "external matrix fast release" T 600 mg po once, followed 48 hours later (Day 11) by "external matrix slow release" T 600 mg once.
  Interventions: Drug: Acyline; Drug: Testosterone
- Finasteride plus Oral Testosterone (Experimental): (Day -2 to Day 12) 1 mg Finasteride PO once daily for 14 days total. (Day 1) Acyline 300 mcg/kg once, followed 24 hours later (Day 2) by "immediate release" T 300 mg po once (as a control), followed 24 hours later (Day 3) by "external matrix fast release" T 300 mg once, followed 24 hours later (Day 4) by "external matrix slow release" T 300 mg once, followed 96 hours later (Day 8) by "immediate release" T 600 mg, followed 24 hours later (Day 9) by "external matrix fast release" T 600 mg po once, followed 48 hours later (Day 11) by "external matrix slow release" T 600 mg once.
  Interventions: Drug: Acyline; Drug: Testosterone; Drug: Finasteride

INTERVENTIONS:
Drug: Acyline — 300 mcg/kg
Drug: Testosterone — 24 hours after acyline administration on Day 2 "immediate release" Testosterone (T) 300 mg po once (as a control), followed 24 hours later (Day 3) by "external matrix fast release" T 300 mg once, followed 24 hours later (Day 4) by "external matrix slow release" T 300 mg once, followed 96 hours later (Day 8) by "immediate release" T 600 mg, followed 24 hours later (Day 9) by "external matrix fast release" T 600 mg po once, followed 48 hours later (Day 11) by "external matrix slow release" T 600 mg once.
  Other Names: Oral Testosterone
Drug: Finasteride — 1 mg PO once daily [day -2 to day 12) 14 days total
  Other Names: Proscar, Propecia, Fincar, Finpecia, Finax, Finast, Finara, Finalo,; Prosteride, Gefina, Appecia, Finasterid IVAX, Finasterid Alternova,; Hyplafin, Penester, Finpros, Tectum, Prezepa
  Arms: Finasteride plus Oral Testosterone

SUMMARY:
We propose a study to determine the single-dose pharmacokinetics of these two novel formulations of testosterone in normal men with experimentally induced hypogonadism.

DETAILED DESCRIPTION:
This is an 2-3 month open-label, two week pharmacokinetic study of two novel formulations of oral testosterone (T), in normal men whose endogenous T production has been temporarily suppressed by the administration of the potent GnRH antagonist Acyline. We will be determining the relative pharmacokinetics of six different oral formulations of T in both rapid and slow release compared to the immediate release preparation studied previously by our group.

ELIGIBILITY:
Inclusion Criteria:

* males between 18 to 50 years of age in good general health based on normal screening evaluation
* must agree not to participate in another research drug study during participation
* must agree to not donate blood during the study
* must be willing to comply with the study protocol and procedures
* must agree to use an acceptable form of contraception
* agrees to not take medications other than the study drugs for the duration of the study

Exclusion Criteria:

* Subject in poor health, determined by medical history physical and lab results
* a known history or current use of alcohol, drug or steroid abuse and/or use of more than 3 alcohol beverages per day
* Participation in a long-term contraceptive study within the past two months
* History of bleeding disorders or current use of anti-coagulants
* History of sleep apnea and/or major psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Plymate SR "Male Hypogonadism" in Principles and Practice of Endocrinology and Metabolism (3rd. Ed). Ed. Kenneth Becker, pp:1125-1150
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Amory JK, Page ST, Bremner WJ. Oral testosterone in oil: pharmacokinetic effects of 5alpha reduction by finasteride or dutasteride and food intake in men. J Androl. 2006 Jan-Feb;27(1):72-8. doi: 10.2164/jandrol.05058. PMID 16400081
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Result] Snyder CN, Clark RV, Caricofe RB, Bush MA, Roth MY, Page ST, Bremner WJ, Amory JK. Pharmacokinetics of 2 novel formulations of modified-release oral testosterone alone and with finasteride in normal men with experimental hypogonadism. J Androl. 2010 Nov-Dec;31(6):527-35. doi: 10.2164/jandrol.109.009746. Epub 2010 Apr 8. PMID 20378927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through news media (newspaper, website) and college campus bulletin boards in Seattle WA, between April 2008-March 2009.
Pre-assignment Details: 19 participants recruited; 19 screened, 2 excluded.
Groups:
- Testosterone Only: (Day 1) Acyline 300 mcg/kg once, followed 24 hours later (Day 2) by "immediate release" T 300 mg po once (as a control), followed 24 hours later (Day 3) by "external matrix fast release" T 300 mg once, followed 24 hours later (Day 4) by "external matrix slow release" T 300 mg once, followed 96 hours later (Day 8) by "immediate release" T 600 mg, followed 24 hours later (Day 9) by "external matrix fast release" T 600 mg po once, followed 48 hours later (Day 11) by "external matrix slow release" T 600 mg once.
- Testosterone Plus Finasteride: (Day -2 to Day 12) 1 mg Finasteride PO once daily for 14 days total. (Day 1) Acyline 300 mcg/kg once, followed 24 hours later (Day 2) by "immediate release" T 300 mg po once (as a control), followed 24 hours later (Day 3) by "external matrix fast release" T 300 mg once, followed 24 hours later (Day 4) by "external matrix slow release" T 300 mg once, followed 96 hours later (Day 8) by "immediate release" T 600 mg, followed 24 hours later (Day 9) by "external matrix fast release" T 600 mg po once, followed 48 hours later (Day 11) by "external matrix slow release" T 600 mg once.
Period: Overall Study
Arm/Group | Testosterone Only | Testosterone Plus Finasteride
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Only | Testosterone Plus Finasteride | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26 (4) | 28 (8) | 27 (4)
Estradiol [Mean (Standard Deviation); unit: pmol/L] | 70.1 (16.1) | 114 (54) | 92.0 (35.0)
Height [Mean (Standard Deviation); unit: centimeters] | 178 (5) | 179 (7) | 178.5 (6)
Sex Hormone Binding Globulin (SHBG) [Mean (Standard Deviation); unit: nmol/L] | 35.5 (12.8) | 32.5 (19.6) | 34 (16.2)
Testosterone (T) [Mean (Standard Deviation); unit: nmol/L] | 14.5 (2.5) | 16.8 (8.9) | 15.65 (5.7)
Weight [Mean (Standard Deviation); unit: kilogram] | 83 (18) | 89 (22) | 86 (20)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve-Serum T
Time Frame: 14 days
Measure: Mean (Standard Error); unit: nmol*h/L
Arm/Group | Testosterone Only | Testosterone Plus Finasteride
Number analyzed (Participants) | 8 | 8
nmol*h/L
  external matrix 'immediate' release | 143 (47) | 198 (86)
  external matrix 'fast' release | 144 (44) | 384 (273)
  external matrix 'slow' release | 162 (60) | 237 (141)
Statistical Analysis 1: Comparison: Testosterone Only vs Testosterone Plus Finasteride; Test type: Non-Inferiority or Equivalence — A sample size of 8 per group was estimated to confer an 80% power to detect a 40% difference in testosterone AUC with a standard deviation of 20% at an alpha of 0.05; p < 0.05, Wilcoxon sign-rank

2. Secondary Outcome: Area Under the Curve-serum DHT
Time Frame: 14-days
Measure: Mean (Standard Error); unit: nmol*h/L
Arm/Group | Testosterone Only | Testosterone Plus Finasteride
Number analyzed (Participants) | 8 | 8
nmol*h/L
  external matrix 'immediate' release | 36 (13) | 23 (10)
  external matrix 'fast' release | 42 (21) | 26 (12)
  external matrix 'slow' release | 39 (16) | 26 (11)
Statistical Analysis 1: Comparison: Testosterone Only vs Testosterone Plus Finasteride; Test type: Non-Inferiority or Equivalence — No power calculation was performed for this pilot study; p < 0.05, Wilcoxon sign-rank

3. Secondary Outcome: Area Under the Curve-E2
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Testosterone Only | Testosterone Plus Finasteride
Number analyzed (Participants) | 8 | 8
nmol*h/L
  external matrix 'immediate' release | 1812 (405) | 2241 (783)
  external matrix 'fast' release | 1961 (528) | 2002 (861)
  external matrix 'slow' release | 1944 (652) | 3129 (1574)
Statistical Analysis 1: Comparison: Testosterone Only vs Testosterone Plus Finasteride; Area-under-the-curve for serum estradiol; Test type: Non-Inferiority or Equivalence — No power calculation was performed for this pilot study; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Testosterone Only | Testosterone Plus Finasteride
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Only (N=8) | Testosterone Plus Finasteride (N=8)
Decreased Libido (Reproductive system and breast disorders) | 1 (2) | 2 (2)
Elevated aspartate aminotransferase (Endocrine disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (7)
Headache (General disorders) | 3 (4) | 3 (3)
Hot flashes (Endocrine disorders) | 2 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes